CLINICAL TRIAL: NCT03986476
Title: The Effect of Two Probiotic Products on the Intestinal Barrier Function in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Robert Brummer, Professor, MD, PhD, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2018/450
Record Dates: First submitted 2019-06-07; First posted 2019-06-14 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: IBS
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactobacillus reuteri strain 1 (Experimental): Probiotic compound
  Interventions: Dietary Supplement: Probiotics
- Lactobacillus reuteri strain 2 (Experimental): Probiotic compound
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — 5x10^8 colony forming units (CFU) of each probiotic strain, two capsules per day over six weeks
  Arms: Lactobacillus reuteri strain 1; Lactobacillus reuteri strain 2
Other: Placebo — Similar in shape and taste to intervention capsules but without the probiotic components, two capsules per day over six weeks
  Arms: Placebo

SUMMARY:
This study will investigate the effects of supplementation with two different probiotic products (Lactobacillus reuteri strains) on the intestinal barrier function, gut health and stress symptoms in diarrhoea-predominant irritable bowel syndrome (IBS-D) patients.

DETAILED DESCRIPTION:
After having given their written informed consent, subjects will complete screening procedures to evaluate their eligibility for the study (visit 1). Study participants will undergo two baseline visits (visits 2 and 3, 3 weeks apart) to account for individual variations, and will then be randomly assigned to 6-week intake of one of two Lactobacillus reuteri strains, or placebo in a ratio of 1:1:1 (stratified by sex). Participants will attend a study visit three weeks into the intervention (visit 4) and at the end of the intervention (visit 5, week 6). The intestinal permeability will be assessed using a standardized multi-sugar test at visit 2, visit 3, visit 4, and at end of intervention (visit 5). Blood, saliva and faecal samples will be collected at visit 2-5. In addition, gastrointestinal symptoms will be recorded at those visits (using Gastrointestinal symptom rating scale-IBS, GSRS-IBS; IBS severity scoring system, IBS- SSS). Quality of life using the 5Q-5D-5L and Hospital Anxiety and Depression Scale (HADS) scores will also be recorded at those visits. In addition, at visit 3 and visit 5, the IBS-Quality of life (IBS-QoL) and the Perceived Stress Scale (PSS) will be completed. In a daily diary, participants will record stool frequency and consistency from visit 2 until end-of-study visit 5. Dietary habits of the patients will be assessed via a food frequency questionnaire (FFQ) and a 3-day food diary before the intervention (between visit 2 and 3).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Fulfilled Rome IV diagnostic criteria for IBS with predominant diarrhoea
* Mild-to-severe IBS symptoms according to the IBS severity scoring system (IBS-SSS; a score of ≥75)
* Age: 18-65 years

Exclusion Criteria:

1. Known organic gastrointestinal disease (e.g. inflammatory bowel disease, IBD)
2. Previous abdominal surgery which might influence gastrointestinal function, except appendectomy and cholecystectomy
3. History of or present gastrointestinal malignancy or polyposis
4. Recently (within the last 6 months) diagnosed gastrointestinal infection
5. Current diagnosis of dementia, severe depression, major psychiatric disorder, or other incapacity for adequate cooperation
6. Chronic neurological/neurodegenerative diseases (e.g. Parkinson's disease, multiple sclerosis)
7. Autoimmune disease and/or patients receiving immunosuppressive medications
8. Chronic pain syndromes (e.g. fibromyalgia)
9. Chronic fatigue syndrome
10. Severe endometriosis
11. Coeliac disease
12. Recently (within the last 3 months) diagnosed lactose intolerance
13. Females who are pregnant or breast-feeding
14. Regular intake of systemic corticosteroids and anti-inflammatory medication (including non-steroidal anti-inflammatory drugs, NSAIDs) during the last 3 months or incidental use in the last 2 weeks prior to randomisation
15. Recent (< 4 weeks) intake of proton pump inhibitors, PPIs (e.g., omeprazol)
16. Use of anti-depressants in the last 3 months
17. Regular oral intake of mast cell stabilising drugs (e.g. sodium cromoglycate) during the last 3 months or incidental use in the last 2 weeks prior to screening
18. Antimicrobial treatment 6 weeks prior to first screening visit
19. Antimicrobial prophylaxis (eg. acne, urinary tract infection)
20. Regular consumption of probiotic products 4 weeks prior to first baseline visit
21. Concurrent or recent (<4 weeks) use of nutritional supplements or herb products affecting intestinal function (e.g. aloe vera, St. John´s Wort, fibres, prebiotics) if the investigator considers those could affect the study outcome.
22. Inability to maintain exercise routine and dietary pattern during the study.
23. Abuse of alcohol or drugs
24. Any clinically significant present or past disease/condition which in the investigator's opinion could interfere with the results of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Change in small intestinal permeability after 6 weeks (urinary lactulose/rhamnose ratio, 0-5h) | 6 weeks
  Difference in small intestinal permeability, measured as the urinary lactulose/rhamnose secretion ratio (0-5h), after a 6-week intervention with the probiotic products compared to the placebo product

SECONDARY OUTCOMES:
Change in small intestinal permeability after 3 weeks (urinary lactulose/rhamnose ratio, 0-5h) | 3 weeks
  Difference in small intestinal permeability, measured as the urinary lactulose/rhamnose secretion ratio (0-5h), after a 3-week intervention with the probiotic products compared to the placebo product
Change in whole gut permeability after 6 weeks (urinary sucralose/erythritol ratio, 0-24h) | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in whole gut permeability, measured as urinary sucralose/erythritol excretion ratio (0-24hrs)
Change in whole gut permeability after 3 weeks (urinary sucralose/erythritol excretion ratio, 0-24h) | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in whole gut permeability, measured as urinary sucralose/erythritol excretion ratio (0-24hrs)
Change in colonic permeability after 6 weeks (urinary sucralose/erythritol ratio, 5-24h) | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in colonic permeability, measured as urinary sucralose/erythritol ratio (5-24hrs)
Change in colonic permeability after 3 weeks (urinary sucralose/erythritol ratio, 5-24hrs) | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in colonic permeability, measured as urinary sucralose/erythritol ratio (5-24hrs)
Change in gastroduodenal permeability after 6 weeks (urinary sucrose excretion, 0-5hrs) | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in gastroduodenal permeability, measured as urinary sucrose excretion (0-5hrs)
Change in gastroduodenal permeability after 3 weeks (urinary sucrose excretion, 0-5hrs) | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in gastroduodenal permeability, measured as urinary sucrose excretion (0-5hrs)
Change in inflammatory status after 3 weeks | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in inflammatory markers in blood (e.g. high-sensitive C-reactive protein)
Change in inflammatory status after 6 weeks | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in inflammatory markers in blood (e.g. high-sensitive C-reactive protein)

OTHER OUTCOMES:
Change in stool frequency and consistency (daily diary on bowel movement using Bristol Stool Chart) | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in stool frequency and consistency
Change in stool frequency and consistency (daily diary on bowel movement using Bristol Stool Chart) | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in stool frequency and consistency
Change in gastrointestinal symptoms measured by the IBS-specific gastrointestinal symptom rating scale (GSRS-IBS) | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in gastrointestinal symptoms (GSRS-IBS total score range 0-3, 0-no symptoms, 3-extreme degree of symptoms)
Change in gastrointestinal symptoms measured by the IBS symptom severity score (IBS-SSS) | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in gastrointestinal symptoms (IBS-SSS, total score range 0-500, 0-no symptoms, 500-extreme degree of symptoms)
Change in gastrointestinal symptoms measured by the IBS-specific gastrointestinal symptom rating scale (GSRS-IBS) | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in gastrointestinal symptoms (GSRS-IBS total score range 0-3, 0-no symptoms, 3-extreme degree of symptoms)
Change in gastrointestinal symptoms measured by the IBS symptom severity score (IBS-SSS) | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in gastrointestinal symptoms (IBS-SSS, total score range 0-500, 0-no symptoms, 500-extreme degree of symptoms)
Change in quality of life measured by IBS-specific quality of life (IBS-QOL) questionnaire | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in quality of life (IBS-QOL total range, range: 0-100, 0-low quality of life, 100-high quality of life)
Change in quality of life measured by IBS-specific quality of life (IBS-QOL) questionnaire | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in quality of life IBS-QOL total range, range: 0-100, 0-low quality of life, 100-high quality of life)
Change in perceived stress using the perceived stress scale (PSS) | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in perceived stress (PSS range 0-40: 0-no stress, 40-high stress)
Change in perceived stress using the perceived stress scale (PSS) | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in perceived stress (PSS range 0-40: 0-no stress, 40-high stress)
Change in anxiety and depression symptoms using the Hospital Anxiety and Depression Scale (HADS) | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in anxiety and depression symptoms (HADS range: 0 to 21 for anxiety and 0 to 21 for depression, 0-low levels, 21 high levels)
Change in anxiety and depression symptoms using the Hospital Anxiety and Depression Scale (HADS) | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in anxiety and depression symptoms (HADS range: 0 to 21 for anxiety and 0 to 21 for depression, 0-low levels, 21 high levels)
Change in salivary cortisol levels | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in salivary cortisol levels
Change in salivary cortisol levels | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in salivary cortisol levels
Change in intestinal microbiota composition (16S rRNA-based next generation sequencing of faecal samples) after probiotic intervention | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in intestinal microbiota composition
Change in intestinal microbiota composition (16S rRNA-based next generation sequencing of faecal samples) after probiotic intervention | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in intestinal microbiota composition
Change in metabolomic profile in faecal samples after probiotic intervention | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in metabolomic profile in faecal samples
Change in metabolomic profile in faecal samples after probiotic intervention | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in metabolomic profile in faecal samples
Change in metabolomic profile in blood samples after probiotic intervention | 3 weeks
  Difference between intervention with the probiotic products compared to the placebo in metabolomic profile in faecal samples
Change in metabolomic profile in blood samples after probiotic intervention | 6 weeks
  Difference between intervention with the probiotic products compared to the placebo in metabolomic profile in faecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared, only data on group level will

REFERENCES:
- [Derived] Konig J, Roca Rubio MF, Forsgard RA, Rode J, Axelsson J, Grompone G, Brummer RJ. The effects of a 6-week intervention with Limosilactobacillus reuteri ATCC PTA 6475 alone and in combination with L. reuteri DSM 17938 on gut barrier function, immune markers, and symptoms in patients with IBS-D-An exploratory RCT. PLoS One. 2024 Nov 1;19(11):e0312464. doi: 10.1371/journal.pone.0312464. eCollection 2024. PMID 39485760